CLINICAL TRIAL: NCT05961228
Title: Back Muscle Function During Exercise With and Without Correction According to the "Schroth" Method in Adolescents With Scoliosis
Brief Title: Back Muscle Function in Adolescents With Idiopathic Scoliosis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Haifa (Other)
Responsible Party: Principal Investigator, Gali Dar, PHD, Prof., University of Haifa
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: 161/23
Record Dates: First submitted 2023-07-18; First posted 2023-07-27 (Actual); Last update posted 2026-01-26 (Actual); Status verified 2026-01

CONDITIONS: Scoliosis Idiopathic; Scoliosis; Adolescence
MeSH Terms: conditions — Scoliosis | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: one group - adolescent with scoliosis. The function and asymmetry of back muscles will be examined in different positions and with specific spinal corrections based on scoliosis pattern and according to the "Schroth method" in the entire sample.
Masking Description: participants will not be aware of the "Schroth method" or the difference between the exercises
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- scoliosis (Other): adolescent age 10-15 with idiopathic scoliosis
  Interventions: Other: exercise

INTERVENTIONS:
Other: exercise — Three different posture with and without correction according to the "Schroth" method

SUMMARY:
The function and asymmetry of back muscles will be examined in different positions and with specific spinal corrections based on scoliosis pattern and according to the "Schroth method" in adolescents with idiopathic scoliosis.

DETAILED DESCRIPTION:
The study aim is to examine function and asymmetry of back muscles in different positions and with and without specific spinal corrections based on scoliosis pattern and according to "Schroth ethod" in adolescenet idiopathic scoliosis. The will include adolescents aged 10-14 years diagnosed on X-ray with idiopathic scoliosis of 15-400 Cobb angle. Participants will undergo an assessment that includes: demographic questionnaire, pain severity measured by the visual analog scale , quality of life questionnaire for patients with scoliosis (SRS-22), Adam's Forward Bend Test, spine rotation angle assessment using a scoliometer, leg length measurement, hip range of motion using goniometer, Risser sign, Coronal trunk balance and Sagittal vertical axis- according to X-ray, scoliosis classification.

Following examination, participants will perform three exercises that activate back muscles in three different positions: supine lying, side lying and standing. Each exercise will be performed twice: the first time without and the second time with specific corrections of the scoliosis. The exercises will be performed according to "Schroth" method implying that the corrections of the spine will be determined according to the scoliosis pattern and classification for the scoliosis (single / double, thoracic, lumbar etc.) and will be conducted via belts, cushions, and bars.

During each exercise, back muscles thickness will be examined and measured via portable diagnostic ultrasound. The muscles will be measured at T7 and L4 levels in resting and contracting positions. Back muscle function will be evaluated by calculating percentage of change between positions rest and contraction position.

Comparison between muscle function with and without correction and correlation of muscle function to quality of life and other morphological parameters will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Adolescents who have been diagnosed by X-ray with idiopathic scoliosis of 15-40°,
* Risser sign zero to four,
* have recent X-rays.

Exclusion Criteria:

* previous back surgery
* have been treated with physical therapy in the past year,

Ages: 10 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 25 (Actual)
Dates: Start 2024-01-10 (Actual); Primary Completion 2025-10-10 (Actual); Study Completion 2025-10-10 (Actual)

PRIMARY OUTCOMES:
Back muscle thickness in centimeters | baseline
  back muscles thickness will be measured in rest and contraction using ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Gali Dar, Prof., Principal Investigator — University of Haifa
Locations (1):
- Haifa University, Department of PHysical Therapy, Haifa, Israel

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: one year following the end of the trial